CLINICAL TRIAL: NCT06530017
Title: A Prospective, Multicenter, Randomized, Double-blind, Parallel Controlled, and Superiority Clinical Trial to Evaluate the Effectiveness and Safety of Ingested, Space Occupying Hydrogel Capsules for Simple Obesity Treatment
Brief Title: Clinical Trial to Evaluate the Ingested, Space Occupying Hydrogel Capsules for Simple Obesity Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IMEIK Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMK-2023-NK001
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Simple Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects in the Study group will be treated with Ingested, Space Occupying hydrogel capsules, which (Experimental): During the treatment period (24 weeks after enrollment), Subjects should take four (4) capsules (Ingested, Space Occupying hydrogel capsules or placebo) with water every day 10~20 minutes before lunch and dinner, and drink at least 500ml of water.
  Interventions: Device: Ingested, Space Occupying hydrogel capsules
- Subjects in the Placebo group will be treated with placebo of the control medical device. (Placebo Comparator): During the treatment period (24 weeks after enrollment), Subjects should take four (4) capsules (Ingested, Space Occupying hydrogel capsules or placebo) with water every day 10~20 minutes before lunch and dinner, and drink at least 500ml of water.
  Interventions: Device: placebo

INTERVENTIONS:
Device: Ingested, Space Occupying hydrogel capsules — During the treatment period (24 weeks after enrollment), Subjects should take four (4) capsules (Ingested, Space Occupying hydrogel capsules or placebo) with water every day 10~20 minutes before lunch and dinner, and drink at least 500ml of water
  Arms: Subjects in the Study group will be treated with Ingested, Space Occupying hydrogel capsules, which
Device: placebo — During the treatment period (24 weeks after enrollment), Subjects should take four (4) capsules (Ingested, Space Occupying hydrogel capsules or placebo) with water every day 10~20 minutes before lunch and dinner, and drink at least 500ml of water
  Arms: Subjects in the Placebo group will be treated with placebo of the control medical device.

SUMMARY:
To evaluate the effectiveness and safety of Ingested, Space Occupying hydrogel capsules for simple obesity treatment

DETAILED DESCRIPTION:
Ingested, Space Occupying hydrogel capsules is indicated to aid in simple obesity treatment with a Body Mass Index (BMI) of 28-40 kg/m2，using under the guidance of a physician.This clinical trial seek to evaluate the efficacy and safety of Ingested, Space Occupying hydrogel capsules for simple obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subjects have a BMI≥28kg/m²and BMI≤40kg/m²

Exclusion Criteria:

* Individuals with secondary obesity, such as hypothyroidism, Cushing's syndrome, etc.
* Those who have undergo surgical method within the past 3 months prior to screening, or plan to lose weight by surgical method during the clinical trial.
* Weight loss exceeding >5% (self-report) within the past 3 months prior to screening.
* Individuals with uncontrolled diabetes mellitus (fasting blood glucose≥7.0mmol/L or glucose loading after 2 hours blood glucose≥11.1mmol/L or glycosylated hemoglobin≥7.0%) .
* Within 1 month before screening or planning to use drugs or health products that may cause significant weight gain or loss during the clinical trials, including biguanides,α-glycosidase inhibitors, SGLT-2 inhibitors, GLP-1 receptor agonists, leptinoid drugs, sympathomimetic drugs, esterase inhibitors, lipolytic injections, sulfonamides, systemic glucocorticoids (more than 1 week), estrogen, thyroid hormones or preparations, antipsychotic or antidepressant drugs, Chinese patent medicines and Chinese herbal medicines, etc.
* Patients with central nervous system diseases (including but not limited to any type of seizures or strokes) and other related neurological diseases or mental illnesses.
* Those who have suffered or are suffering from swallowing disorders, gastroesophageal reflux disease, gastric or duodenal ulcers, gastroparesis, esophageal and gastric varices, intestinal obstruction or suspected small bowel adhesions, pyloric obstruction, Crohn's disease, ulcerative colitis and other diseases, acute/chronic pancreatitis, as well as a history of gastrointestinal surgery (except those related to appendectomy and intestinal polypectomy), abdominal radiation therapy, and gastrointestinal bleeding.
* Those who have AIDS or a history of cancer within the past 5 years.
* Patients with poorly controlled hypertension, i.e., systolic blood pressure (SBP) > 165mmHg and/or diastolic blood pressure (DBP) >95mmHg.
* Patients with renal insufficiency, i.e., estimated glomerular filtration rate (eGFR<30 ml/min/1.73m2)* calculated by the CKD-EPI creatinine equation as defined by the KDIGO 2012 classification.
* Patients with impaired liver function, that is, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal, or total bilirubin (TBIL) > 3 times the upper limit of normal.
* Those who stop smoking within the past 6 months before the screening period or consider stop smoking during the trial.
* Those who have planned surgery in the past 6 months.
* Pregnant or breastfeeding, planning to become pregnant during the trial (or males unwilling to use an adequate method of contraception), or having a positive pregnancy test result during the screening period.
* Individuals with a history of allergies to cellulose, titanium dioxide, citrate acid and succinic acid.
* Those with severe cardiovascular and cerebrovascular diseases or systemic failure that affects treatment.
* The investigator judges that the subject has other systemic diseases that are not suitable for participating in this trial, and the abnormal laboratory test results are determined by the investigator whether they can be enrolled.
* Participated in clinical trials of other drugs or medical devices within 30 days prior to the screening period.
* Other circumstances that the investigator deems inappropriate to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight loss percentage from baseline at Week 24 | 24 weeks
  Calculation formula:Weight loss percentage from baseline = (weight at Week 24 after enrollment of subject - baseline weight) / baseline weight×100%
Response rate of weight loss at week 24 after enrollment | 24 weeks
  Calculation formula:Weight loss response rate = Number of subjects with ≥5% weight loss percentage from baseline/total number of subjects ×100%.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Li, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (10):
- China (10):
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third XiangYa Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Luoyang
  - QILU Hospital Of Shandong University, Jinan, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality